CLINICAL TRIAL: NCT06928363
Title: A First-in-human, Multicenter, Open-label Phase I/II Investigational Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of KY-0301 as Monotherapy in Patients With Advanced Solid Tumors.
Brief Title: A First-in-human Study of KY-0301 in Patients With Advanced Solid Tumors.
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novatim Immune Therapeutics (Zhejiang) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KY-0301-XG101
Record Dates: First submitted 2025-03-31; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-03

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Dose escalation/Expansion：KY-0301 (Experimental): KY-0301, 0.3 mg/kg~ 2.0 mg/kg.i.v. Q2W，4 weeks/cycle
  Interventions: Drug: KY-0301
- Cohort A:EGFRm NSCLC (Experimental): KY-0301, .i.v. Q2W，4 weeks/cycle
  Interventions: Drug: KY-0301
- Cohort B:EGFRwt NSCLC (Experimental): KY-0301, 0.3 mg/kg~ 2.0 mg/kg.i.v. Q2W，4 weeks/cycle
  Interventions: Drug: KY-0301
- Cohort C:CRC (Experimental): KY-0301, 0.3 mg/kg~ 2.0 mg/kg.i.v. Q2W，4 weeks/cycle
  Interventions: Drug: KY-0301
- Cohort D: other solid tumor (Experimental): KY-0301, 0.3 mg/kg~ 2.0 mg/kg.i.v. Q2W，4 weeks/cycle
  Interventions: Drug: KY-0301

INTERVENTIONS:
Drug: KY-0301 — KY-0301 is an antibody-drug conjugate (ADC) targeting both EGFR and c-Met, developed independently by Novatim Immune Therapeutics (Zhejiang) Co., Ltd

SUMMARY:
This trial is a first-in-human, multicenter, open-label Phase I/II clinical study to evaluate the safety, tolerability, pharmacokinetics, and preliminary efficacy of KY-0301 as monotherapy in patients with advanced solid tumors. This trial will be conducted at approximately multi-sites nationwide, and approximately110~212 participants with unresectable locally advanced or metastatic solid tumors will be invited to participate. The study consists of three parts: Phase I dose escalation & dose expansion phases of KY-0301 as monotherapy, Phase II cohort expansion phase of KY-0301 as monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Know the trial information before the start of the study and voluntarily sign an informed consent form (ICF).
* Aged ≥ 18 years, male or female.
* Agree to follow and be capable of completing all study procedures.
* Female weight > 45 kg, male weight > 50 kg, with a BMI ≥18 kg/m2
* Tumor Types:

Part I, Patients with histologically or cytologically confirmed locally advanced or metastatic solid tumors; Patients who have failed existing standard treatment regimens, are intolerant to standard treatment, have no standard treatment regimen, or are currently not suitable for standard treatment.

Part II, Cohort A: Histologically or cytologically confirmed locally advanced or metastatic non-squamous non-small cell lung cancer (NSCLC) ;Patients who have previously received EGFR TKI and at least 1st line platinum-containing two-drug standard systemic chemotherapy; Patients must have radiographically confirmed disease progression from the last prior anticancer therapy to the enrollment in this study. Cohort B: Histologically or cytologically confirmed NSCLC with no actionable genetic mutations have been identified ；have received at least first-line anti-PD - (L) 1 immunotherapy and chemotherapy . Cohort C :Histologically or cytologically confirmed CRC; Patients who have previously received SoC; chemotherapy above the 3rd line is received in the systemic treatment phase. Cohort D: other histologically or cytologically confirmed locally advanced or metastatic solid tumors

Exclusion Criteria:

* History of intolerance to ADC therapy composed of monomethyl auristatin E (MMAE).
* Inadequate washout period of prior antitumor therapy prior to the first dose
* Patients who have undergone major surgery (excluding diagnostic surgery) within 4 weeks prior to first dose or those who plan to undergo major surgery during the study period. Interventional or ablative procedures for tumor treatment within 2 weeks prior to the first dose of the investigational drug.
* Previous allogeneic bone marrow transplantation or previous solid organ transplantation.
* Systemic steroid use (>20 mg/day of prednisone or equivalent) or other immunosuppressive treatments within 2 weeks prior to first dose of the investigational drug, with the following exceptions: Intranasal, inhaled, or local steroid injections (e.g., intra-articular injections); Physiologic doses of systemic steroids as replacement therapy (e.g., physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency);Use of steroids to prevent hypersensitivity reactions or to prevent antiemetic (e.g., computed tomography (CT) prophylaxis).
* Received any live vaccine within 4 weeks prior to the first dose or plan to receive a live vaccine during the study.
* History of leptomeningeal carcinomatosis or carcinomatous meningitis.
* Brain metastasis or spinal cord compression, except for Patients with asymptomatic brain metastases
* Uncontrolled or clinically significant cardiovascular or cerebrovascular diseases
* Clinically significant concomitant pulmonary diseases
* Patients with symptomatic or unstable third-spacing (e.g., pleural effusion, ascites, pericardial effusion) require repeated drainage.
* History of gastrointestinal perforation and/or fistula within 6 months prior to the first dose, or the presence of active gastric ulcer, duodenal ulcer, ulcerative colitis, gastrointestinal obstruction, or any other gastrointestinal disease that the investigator deems may cause bleeding or perforation.
* Patients with severe infection [≥ Grade 3 per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0] prior to first dose
* Patients with HIV infection or those who test positive for syphilis antibodies with a positive titer test.
* Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection. Active HBV is defined as positive hepatitis B surface antigen (HBsAg) and/or positive hepatitis B core antibody (HBcAb), with HBV DNA levels above the detectable lower limit of the study site; active HCV is defined as positive hepatitis C antibodies with HCV RNA levels above the detectable lower limit of the study site.
* Non remission of toxicity from previous anticancer therapy is defined as non remission of toxicity (other than alopecia and pigmentation) to NCI CTCAE v5.0 ≤ Grade 1, baseline, or inclusion/exclusion criteria. Patients with chronic Grade 2 toxicities may be eligible for enrollment if the toxicity is asymptomatic or adequately controlled with stable medication, after discussion with the sponsor.
* History of severe allergic reactions to drugs
* Any other primary malignancy within 5 years prior to first dose of the investigational drug, except for low-risk tumors such as adequately resected basal cell skin cancer, cervical carcinoma in situ, or papillary thyroid carcinoma .etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-11-12 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Occurrence of dose-limiting toxicity (DLT) | 28 days
  DLT is defined as an adverse event (AE) that meets protocol defined DLT criteria during cycle 1 and is at least possibly related to study drug.
MTD | Up to 24 Months
  The maximum tolerated dose (MTD) is defined as the maximum dose where the number of cases of DLT ≤ 1/6 of the total number of cases during the DLT observation period. At least 6 evaluable subjects are required to determine MTD.

SECONDARY OUTCOMES:
The area under curve (AUC) of KY-0301 (ADC) in plasma | Up to 24 Months
  Area under the plasma concentration versus time curve
The immunogenicity of KY-0301 | Up to 24 Months
  Occurrence of anti-drug antibodies (ADA)
Objective response rate (ORR) | Up to 24 Months
  defined as percentage of participants with confirmed best overall response of confirmed partial response (PR) or better per investigator review according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Progression-free survival (PFS) | Up to 24 Months
  PFS is defined as time from first study treatment to a documented disease progression according to RECIST, version 1.1, as determined by the investigator, or death due to any cause, whichever occurs earlier.
The maximum concentration (Cmax) of KY-0301 in plasma | up to 24 months
  The Peak Plasma Concentration of KY-0301 in plasma

IPD SHARING:
Plan to Share IPD: No